CLINICAL TRIAL: NCT03776500
Title: Safety, Tolerability and Pharmacokinetic Profile of PBTZ169 Formulated as Native Crystal Powder: Multiple Ascending Doses, Randomized, Placebo- Controlled, Parallel-group, Sequential Phase Ib Trial in Healthy Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability and Pharmacokinetics of PBTZ169 in Multiple Dosing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovative Medicines for Tuberculosis (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IM-006-13
Record Dates: First submitted 2018-12-13; First posted 2018-12-14 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — macozinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Panel A - Active (Experimental): N = 6, 150 mg twice daily of PBTZ169
  Interventions: Drug: PBTZ169
- Panel A - Placebo (Placebo Comparator): N = 2, 150 mg twice daily of PBTZ169 matching placebo
  Interventions: Drug: Placebo
- Panel B - Active (Experimental): N = 6, 300 mg twice daily of PBTZ169
  Interventions: Drug: PBTZ169
- Panel B - Placebo (Placebo Comparator): N = 2, 300 mg twice daily of PBTZ169 matching placebo
  Interventions: Drug: Placebo
- Panel C - Active (Experimental): N = 6, 600 mg once daily of PBTZ169
  Interventions: Drug: PBTZ169
- Panel C - Placebo (Placebo Comparator): N = 2, 600 mg once daily of PBTZ169 matching placebo
  Interventions: Drug: Placebo
- Panel D - Active (Experimental): N = 6, 600 mg twice daily of PBTZ169
  Interventions: Drug: PBTZ169
- Panel D - Placebo (Placebo Comparator): N = 2, 600 mg twice daily of PBTZ169 matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBTZ169 — PBTZ169 crystalline supplied as powder for oral solution
  Arms: Panel A - Active; Panel B - Active; Panel C - Active; Panel D - Active
Drug: Placebo — matching placebo supplied as powder for oral solution
  Arms: Panel A - Placebo; Panel B - Placebo; Panel C - Placebo; Panel D - Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multiple ascending dose study conducted at one study center in Switzerland.

Four (4) panels (A, B, C and D) of 8 male subjects (6 active and 2 placebo) each receiving multiple doses of PBTZ169 or a matching placebo, at increasing dose levels, once or twice daily.

Subjects will participate in only one panel. Blocks of 4 subjects (3 under active treatment, 1 under placebo) will be investigated in parallel. Panels will start sequentially.

Safety will be assessed throughout the study; serial ECGs and serial blood samples will be collected for the safety and PK assessment of PBTZ169.

Dose escalation will be allowed once the Trial Safety Board has determined that adequate safety and tolerability after each panel completion has been demonstrated to permit proceeding to the next panel.

In addition, a preliminary assessment of the drug interaction potential of PBTZ169 will be done by the measurement of inhibition or induction of human cytochromes through the metabolism of microdoses of standard probe substrates

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged between 18 and 48 years
* Body weight (BW) ranging between 55 and 95 kg, providing body mass index (BMI) is between 18 and 28 kg/m2
* Absence of significant findings in the medical history and physical examination as judged by the Investigator, especially for cardiovascular, pulmonary, haematological and nervous systems
* Absence of significant laboratory abnormalities as judged by the Investigator. Gilbert's syndrome (increased total and unconjugated bilirubin when fasting) will be accepted if mild. Moderate creatine kinase increases (up to 600 IU/L) without clinical abnormalities, commonly found in physically active young males.
* Absence of clinically significant abnormalities on 12-lead ECG
* Negative urine drug screen (amphetamines, benzodiazepines, cannabis, cocaine, opiates)
* Commitment to refrain from travel outside Europe over the whole study duration
* Ability to understand the procedures, agreement to participate and willingness to give written informed consent
* Co-operative attitude and availability for scheduled visits over the entire study period
* Commitment to refrain from alcohol and tobacco consumption over the whole study period.

Exclusion Criteria:

* History of major cardiovascular, pulmonary, hepatic, immunological, renal, haematological, gastrointestinal, genitourinary, neurological, or rheumatologic disorders
* Active diseases of any type, including inflammatory disorders and infections. Mild acne is permissible providing no systemic or local treatment is provided or planned (except for cleaning lotions)
* History of significant allergy or asthma. Allergic rhinitis or conjunctivitis is acceptable if non-symptomatic when starting the study and if symptoms are not anticipated to occur during the study to a point that would require corticosteroid therapy (e.g. in case of annual use)
* History of cardiovascular dysfunction if considered as clinically relevant (conduction abnormality, arrhythmia, bradycardia, angina pectoris, cardiac hypertrophy unless elicited by training, pulmonary embolism)
* Hypertension defined as supine blood pressure >150/90 mmHg or recurrent hypotensive events considered as clinically relevant or documented orthostatic hypotension
* Sick sinus syndrome, known long QT syndrome, reproducible observation of corrected QT interval QTc ≥440 msec or of pronounced sinus bradycardia (<40 bpm/min)
* Intense sport activities. Moderate sport is acceptable and activities should remain fairly constant throughout the study
* Any clinically significant laboratory values on screening that are not within normal range on single repeat (Gilbert's syndrome or CK elevations usually acceptable if moderate)
* Positive hepatitis B and C antigen screen
* Positive HIV antibody screen or screen not performed
* Any recent acute illness or sequelae thereof which could expose the subject to a higher risk or might confound the results of the study, according to the evaluation of the investigator
* Treatment in the previous three months with any drug known to have well-defined potential for toxicity to a major organ
* History of hypersensitivity to any drug if considered as serious
* Use of any medication the week prior to study or as based on the 5 plasma half-life rule and throughout study, including aspirin or other over-the-counter (OTC) preparations. Paracetamol is permissible before and during the study as a rescue medication but only with Investigator's permission
* Participation in a clinical investigation or blood donation of 500 ml within the past 3 months
* History of relevant alcohol or drug abuse
* Usual smoking during the last month before participation in the study. Consumption of ≤5 cigarettes/day or equivalent is acceptable providing the subject can totally refrain from smoking from one week before and during the whole study duration
* Usual consumption of a large quantity of coffee, tea, chocolate (more than 4 cups/day) or equivalent (Cola drinks), during the last month before participation in the study
* Current regular (i.e. 3 times per week or more) consumption of large quantities of alcohol or wine (>0.5 L wine/day) or equivalent (i.e. more than 50 g ethanol per day), during the last month before participation in the study. Alcohol is not allowed during the whole study period
* Project to conceive a child during the study period (by principle of precaution, while no indication exists for a definite reproductive risk following paternal exposure)
* Psychological status which could impact on the subject's ability to give informed consent
* Any feature of the subject's medical history or present condition which, in the Investigator's opinion, could confound the results of the study, complicate its interpretation, or represent a potential risk for the subject.

Ages: 18 Years to 48 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of increasing multiple oral doses of PBTZ169 in healthy male adult subjects evaluated by Treatment Emergent Adverse Events (TEAEs). | Days 0-17
  Evaluation by thorough monitoring of Treatment Emergent Adverse Events (TEAEs) following doses of PBTZ169 crystalline or placebo

SECONDARY OUTCOMES:
Relative oral bioavailability assessment of PBTZ169 in healthy male subjects after multiple dosing | Days 0-17
  Estimation from the ratio of area under plasma concentration curves (AUCs) determined after the administration of PBTZ169
Pharmacokinetics (PK) of multiple oral doses of PBTZ169 using Cmax | Days 0-17
  Determination of non-compartmental PK parameter Maximum Plasma Concentration [Cmax] after determination of the amount of the parent compound and its known metabolites in plasma samples
Pharmacokinetics (PK) of multiple oral doses of PBTZ169 using Tmax | Days 0-17
  Determination of non-compartmental PK parameter Time of maximum observed Plasma Concentration [Tmax] after determination of the amount of the parent compound and its known metabolites in plasma samples
Metabolism interaction of multiple oral doses of PBTZ169 by measuring ratios of 7 probe substrates before the first and and after the last dose | Days -1 to 14
  Measurement of the ratios of 7 probe of known substrates of human Cytochome P-450 enzyme family before the first and and after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Stewart T Cole, Prof, Study Chair — innovative Medicines for Tuberculosis (iM4TB)
Locations (1):
- Division of Clinical Pharmacology, Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland